CLINICAL TRIAL: NCT07364929
Title: Altered Non-Visual Photoreception in Patients With Glaucoma: Impacts on Sleep, Alertness, Mood, and Cognition
Acronym: EyeQ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Singapore National Eye Centre (Other Government); Singapore Eye Research Institute (Other); National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Raymond P. Najjar, PhD, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: DSRB 2024/00123
Record Dates: First submitted 2025-12-16; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Glaucoma
Keywords: light; glaucoma; brain; sleep; mood; cognition; alertness
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: In this study, the cross-over model refers to the way each participant experiences both lighting conditions (control light and intervention light). Each participant (whether patient or healthy control) takes part in two experimental sessions during their laboratory visit:
  1. Standard Indoor Light (Control) Condition (~300 lux)
  2. Full-spectrum (Intervention) Condition (~1000 lux) The order of exposure is randomized. Half of the participants start with the standard light, then switch to the full-spectrum light. The other half experience the reverse order.
  This randomization prevents order or carryover effects (for example, participants simply performing better the second time because of practice or worse because of fatigue).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with glaucoma (Experimental): Patients undergoing both control and intervention light exposure in a cross-over randomized design.
  Interventions: Other: Full-spectrum light exposure; Other: Standard indoor light exposure (Control)
- Controls (healthy adults) (Active Comparator): Healthy adults following the same procedures compared to patients with glaucoma
  Interventions: Other: Full-spectrum light exposure; Other: Standard indoor light exposure (Control)

INTERVENTIONS:
Other: Full-spectrum light exposure — Participants will be exposed to a full-spectrum white light designed to replicate the spectral quality of natural daylight while maintaining safe, indoor intensity levels. The light source delivers an illuminance of approximately 1000 lux and is free of ultraviolet and infrared wavelengths. Each participant will undergo two periods of light exposure, intermittently, during the laboratory visit at the Eye N' Brain Research Platform (NUS).
  Other Names: Sun-like light
Other: Standard indoor light exposure (Control) — Participants will be exposed to a standard indoor light with an illuminance of approximately 300 lux. Each participant will undergo two periods of light exposure, intermittently, during the laboratory visit at the Eye N' Brain Research Platform (NUS).

SUMMARY:
The goal of this study is to understand how light sensitivity in the eye affects sleep, mood, alertness, and cognition in adults with glaucoma compared to healthy individuals aged 45-75 years.

The main questions it aims to answer are:

1. Do patients with glaucoma experience poorer sleep, mood, alertness, and cognitive function than age-matched healthy adults?
2. Are these changes related to reduced light sensitivity in special retinal cells called intrinsically photosensitive retinal ganglion cells (ipRGCs), lost in glaucoma?
3. Can exposure to safe, full-spectrum indoor light help improve these functions?

Researchers will compare patients with glaucoma and age-matched healthy controls to see if differences in light sensitivity can explain changes in non-visual light responses (i.e., sleep, mood, alertness, and cognition) and whether full-spectrum light exposure can enhance alertness and wellbeing.

Participants will:

1. Complete eye exams and baseline questionnaires about their sleep, daytime sleepiness, mood, and wellbeing.
2. Wear a wrist-worn device for 8-16 days to record their sleep patterns and light exposure.
3. Visit the laboratory for cognitive and attention tests following exposure to two lighting conditions (randomized, cross-over):

   * Standard indoor light (~300 lux)
   * Full-spectrum light (~1000 lux)

This study will help researchers understand how glaucoma affects the brain beyond vision and explore whether light-based interventions can improve quality of life for people living with glaucoma.

DETAILED DESCRIPTION:
Glaucoma is a chronic eye disease that damages retinal ganglion cells (RGCs), leading to progressive loss of vision. Recent evidence suggests that glaucoma may also affect a special subset of RGCs called intrinsically photosensitive retinal ganglion cells (ipRGCs), which contain the light-sensitive pigment melanopsin. These cells are critical for regulating non-visual responses to light, such as sleep, mood, alertness, and cognition, by sending light signals from the eye to various regions of the brain.

Patients with glaucoma often report sleep disturbances, fatigue, and mood changes, yet the biological mechanisms behind these symptoms are not fully understood. It remains unclear whether such non-visual effects result from damage to ipRGCs or from other disease-related factors. Understanding this relationship is important for improving the overall wellbeing and quality of life of individuals living with glaucoma.

This study will therefore investigate how glaucoma affects non-visual responses to light and whether brief, safe exposure to full-spectrum light can improve alertness, sleepiness, and mood. The study combines observational and interventional components to comprehensively assess the link between light perception, brain function, and behavior in glaucoma.

Study Design and Procedures

A total of 120 participants will take part in the study:

1. 60 patients with bilateral primary open-angle glaucoma
2. 60 healthy control participants matched for age (45-75 years)

Each participant attends two study visits:

Visit 1 is done at the clinics (National University Hospital / Singapore National Eye Center) and covers the following:

* Comprehensive eye examination including visual field testing, optical coherence tomography (OCT), fundus photography, autorefraction, visual acuity, color vision, slit-lamp examination and intraocular pressure measurement.
* Evaluation of sleep quality, daytime sleepiness, and mood using validated questionnaires (Pittsburgh Sleep Quality Index (PSQI), Epworth Sleepiness Scale (ESS), and Patient Health Questionnaire (PHQ-9)).
* Assessment of cognitive function (Montreal Cognitive Assessment).
* Measurement of non-visual light sensitivity using handheld chromatic pupillometry, a non-invasive test that evaluates ipRGC function through pupillary light responses.

Participants are given a wrist-worn actigraphy device to record their daily sleep-wake cycles and light exposure for 8-16 days at home, along with a sleep diary.

Visit 2 is done at the laboratory (National University of Singapore - Eye N' Brain Research Platform). After completing actigraphy, participants return for detailed testing of attention, cognition, and vigilance following exposure to two lighting conditions:

1. Control Light Condition: standard indoor lighting (~300 lux)
2. Experimental Light Condition: full-spectrum white light (~1000 lux), designed to mimic the spectral quality of daylight without ultraviolet or infrared radiation.

Participants undergo two sessions of exposure to each of these lights (separated by a period of standard light during which they perform different versions of the MoCA test).

The timing of the visit is individualized based on each participant's sleep/wake cycle. Participants go through the sessions in a cross-over manner and the order of lighting conditions will be randomized to control for order effects.

Following light exposure, the following cognitive tasks are employed while doing eye tracking and cognitive pupillometry:

1. Auditory Psychomotor Vigilance Task (aPVT) to assess alertness or sustained attention
2. Auditory Oddball Task to assess selective attention
3. Time Estimation Task to assess sleepiness objectively
4. Balloon Analogue Risk Task (BART) to assess risk taking behavior
5. Digit Symbol Substitution Task (DSST) to evaluate processing speed and executive function
6. Cognitive pupillometry in response to different shapes.

Subjective rating scales of mood, wellbeing, and sleepiness are administered before and after each lighting condition and after cognitive assessment to monitor fluctuations throughout the session.

ELIGIBILITY:
Inclusion Criteria:

* Patients with glaucoma must meet all of the inclusion criteria to participate in this study.

  * Patients diagnosed with primary open-angle glaucoma (POAG), as indicated by Humphrey Visual Field (HVF) mean deviation (VFMD) scores better than -12 dB in at least one eye during their most recent clinic visit.
  * Patients having spared central vision.
  * Patients aged 45 to 75 years old.
  * Patients with a best-corrected visual acuity better than 6/12
  * English-speaking patients

Healthy controls must meet all of the inclusion criteria to participate in this study:

* Participants aged 50 to 70 years old.
* Participants with a best-corrected visual acuity better than 6/12
* Normal ophthalmic examination
* English-speaking participants

Exclusion Criteria:

* All subjects (patients and controls) meeting any of the exclusion criteria at baseline will be excluded from participation:

  * Participants with myopia exhibiting a refractive error exceeding -8.00 diopters (D)
  * Participants with a history of complicated previous intraocular surgery
  * Participants taking alpha-adrenergic agonist eye drops or other systemic medications or drugs that could affect the pupillary response
  * Participants with any past or current ocular condition (i.e., age-related retinal diseases (e.g., age-related macular degeneration), retinal pigment epithelium diseases (e.g., Best's disease), diabetic retinopathy, or other optic or generalized neuropathies, significant ocular trauma, or any eye condition affecting fixation (eg. Nystagmus)).
  * Participants diagnosed with cataracts at NS3+ (Nuclear Sclerosis) and above, as well as those with Posterior Subcapsular (PSC) cataracts
  * Participants with clinically diagnosed psychiatric or neurologic disorders, including cognitive impairment or dementia
  * Participants with diagnosed mood disorders
  * Participants engaged in night shift work within the past three months, are currently using sleeping pills, or have recently travelled across timezones within a month prior to the study
  * Participants with obstructive sleep apnea
  * Participants with abnormal auditory function
  * Participants with impaired color vision
  * Pre-menopausal women (last menstrual period < 1 year) (If applicable)
  * Patients having unilateral glaucoma, congenital glaucoma, non-glaucomatous optic neuropathy, abnormal central vision
  * Diabetics on treatment

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Subjective Sleep Quality | Baseline (Visit 1)
  Sleep quality is assessed using the Pittsburgh Sleep Quality Index (PSQI), a validated self-report questionnaire measuring subjective sleep quality, sleep latency, duration, efficiency, disturbances, use of sleep medication, and daytime dysfunction over the past month. Higher scores indicate poorer sleep quality.
Subjective Daytime Sleepiness | Baseline (Visit 1)
  Daytime sleepiness is assessed using the Epworth Sleepiness Scale (ESS), a validated questionnaire evaluating the likelihood of dozing in common daytime situations. Higher scores indicate greater daytime sleepiness.
Depressive Symptoms | Baseline (Visit 1)
  Depressive symptoms will be assessed using the Patient Health Questionnaire-9 (PHQ-9), a validated self-report questionnaire measuring the frequency and severity of depressive symptoms over the past two weeks. Higher scores indicate greater depressive symptom severity.
Global Cognitive Function | Baseline (Visit 1)
  Global cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA), a standardized screening tool evaluating executive function, attention, memory, language, and visuospatial abilities.
Global Cognitive Function during light exposure | Immediately after the procedure
  Global cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA), a standardized screening tool evaluating executive function, attention, memory, language, and visuospatial abilities. Alternate validated versions will be used across visits to minimize learning effects.
Median Reaction Time | Immediately after the procedure
  Median reaction time will be assessed using a laboratory-based auditory Psychomotor Vigilance Task (aPVT). Participants will respond to auditory stimuli presented via headphones by pressing a key on a keyboard while viewing a fixation display on a monitor. Reaction time is defined as the interval between stimulus onset and the participant's button press. The primary outcome measure is the median reaction time calculated across all valid trials within the task.
Vigilance Lapses | Immediately after the procedure
  Vigilance lapses will be assessed using a laboratory-based auditory Psychomotor Vigilance Task (aPVT). Participants will respond to auditory stimuli presented via headphones by pressing a key on a keyboard while viewing a fixation display on a monitor. Omission lapses are defined as trials in which no response is registered within the predefined response window following stimulus onset. The outcome measure is the total number of omission lapses across all valid trials.
Long Reation Time Lapses | Immediately after the procedure
  Long reaction time lapses will be assessed using a laboratory-based auditory Psychomotor Vigilance Task (aPVT). Participants respond to auditory stimuli by pressing a key on a keyboard. A long reaction time lapse is defined as any trial in which the reaction time exceeds two times the participant's median reaction time for the task. The outcome measure is the total number of long reaction time lapses across all valid trials.
Anticipatory Responses | Immediately after the procedure
  Anticipatory responses will be assessed using a laboratory-based auditory Psychomotor Vigilance Task (aPVT). Participants respond to auditory stimuli by pressing a key on a keyboard. An anticipatory response is defined as a button press occurring before stimulus onset, reflecting premature responding. The outcome measure is the total number of anticipatory responses across all valid trials.
Sustained Attention Variability | Immediately after the procedure
  Additional reaction time metrics will be derived from the auditory Psychomotor Vigilance Task (aPVT) to characterize response speed distribution and variability. These metrics include reaction time slope across trials, fastest reaction times (e.g., fastest 10%), slowest reaction times (e.g., slowest 10%), and measures of intra-individual reaction time variability. These outcomes provide complementary information on vigilance stability and performance dynamics beyond central tendency measures.
Associative Learning | Immediately after the procedure
  Associative Learning is assessed using a computerized variant of the Digital Symbol Substitution Task (DSST). Associative learning is quantifies by the proportion of correct responses across all trials (accuracy).
Processing Speed | Immediately after the procedure
  Processing speed is assessed using a computerized variant of the Digital Symbol Substitution Task (DSST). Processing speed is quantifies by the median reaction time taken across trials to judge if the presented combination is correct or incorrect (button press).
Visual Attention Allocation | Immediately after the procedure
  Visual attention allocation during the Digit Symbol Substitution Task (DSST) is assessed using eye tracking. Predefined areas of interest (AOIs), including the reference symbol-number set and the presented test pair, will be used to quantify visual strategy. Outcome measures include the number and sequence of visits to each AOI and the proportion of viewing time spent within each AOI across valid trials.
Eye-Movement Behavior | Immediately after the procedure
  Eye-movement behavior during the Digital Symbol Substitution Task (DSST) will be assessed using video-based eye tracking. Metrics will characterize visual exploration and oculomotor behavior and include fixation count and duration, saccade frequency and amplitude, and related summary measures averaged across valid trials.
Selective Attention | Immediately after the procedure
  Cognitive processing of infrequent auditory stimuli will be assessed using a laboratory-based auditory oddball task. Auditory tones will be presented via headphones while participants view a fixation display on a monitor and respond using a keyboard. Accuracy is defined as the proportion of correctly detected target tones and correctly ignored non-target tones across all trials.
Auditory Discrimination Performance | Immediately after the procedure
  Auditory discrimination performance will be assessed using an auditory oddball task. Sensitivity (d') will be calculated based on hit rates (correct detection of target tones) and false alarm rates (responses to non-target tones). Higher d' values indicate greater ability to discriminate infrequent target tones from frequent non-target tones.
Task-Evoked Pupillary Responses | Immediately after the procedure
  Task-evoked pupillary responses will be recorded during performance of the auditory Psychomotor Vigilance Task (aPVT) as well as the oddball task using eye-tracking pupillometry. Changes in pupil size measured during task performance, following stimulus presentation and participant response, will be quantified as indicators of cognitive effort and alertness. Outcome measures include pupil dilation amplitude and response dynamics averaged across valid trials.
Pupillary Responses to Shapes | Immediately after the procedure
  Changes in pupil size during image presentation will be quantified as physiological correlates of the perceived features of a shape, independent of physical luminance.
Objective sleepiness | Immediately after the procedure
  Objective sleepiness will be assessed using a computerized time estimation task. Participants will be instructed to press a button when they believe that a specified time interval has elapsed (10 seconds, 20 seconds, 30 seconds, 60 seconds, and 120 seconds). Time estimation accuracy will be quantified as the difference between the estimated and actual interval duration across trials.
Risk Taking Behavior | Immediately after the procedure
  Risk-taking behavior is assessed using the Balloon Analogue Risk Task (BART), a computerized decision-making task. Adjusted average pumps is calculated as the mean number of pumps on balloons that do not burst (i.e., excluding balloons that explode), providing an index of risk-taking propensity.
Subjective Sleepiness, Mood, and Wellbeing | Immediately after the procedure
  Change in subjective sleepiness, mood, and wellbeing assessed using the Stanford Sleepiness Scale (SSS) and Likert scales before each light exposure (baseline), immediately after exposure (acute effect), and following cognitive assessments (sustained effect).
Sleep Quantity | 8-16 days in between the visits
  Night time sleep quantity (minutes) will be collected through actigraphy watches given to participants.
Sleep Efficiency | 8-16 days between the visits
  Night time sleep efficiency (%) calculated as the amount of time spent asleep (in minutes) by the total amount of time in bed (in minutes) will be measured using actigraphy watches given to participants.
Phasic Pupil Constriction to Blue Light | Baseline (Visit 1)
  Phasic pupil constriction to blue light will be quantified using chromatic pupillometry with a handheld chromatic pupillometer. Phasic pupil constriction to blue light refers to the rapid, transient decrease in pupil diameter that occurs immediately after the onset of a blue light stimulus. It is calculated as a percentage change from baseline.
Phasic Pupil Constriction to Red Light | Baseline (Visit 1)
  Phasic pupil constriction to red light will be quantified using chromatic pupillometry with a handheld chromatic pupillometer. Phasic pupil constriction to red light refers to the rapid, transient decrease in pupil diameter that occurs immediately after the onset of a red light stimulus. It is calculated as a percentage change from baseline.
Maximum Pupil Constriction to Blue Light | Baseline (Visit 1)
  Maximum pupil constriction to blue light will be quantified using chromatic pupillometry with a handheld chromatic pupillometer. Maximum pupil constriction to blue light refers to the greatest reduction in pupil diameter observed following the onset of a blue light stimulus. It is calculated as a percentage change from baseline.
Maximum Pupil Constriction to Red Light | Baseline (Visit 1)
  Maximum pupil constriction to red light will be quantified using chromatic pupillometry with a handheld chromatic pupillometer. Maximum pupil constriction to red light refers to the greatest reduction in pupil diameter observed following the onset of a red light stimulus. It is calculated as a percentage change from baseline.
Pupil Constriction Latency to Blue Light | Baseline (Visit 1)
  Maximum pupil constriction to blue light will be quantified using chromatic pupillometry with a handheld chromatic pupillometer. Constriction latency is defined as the time from blue light onset to the first detectable decrease in pupil diameter relative to baseline. It is measured in seconds.
Pupil Constriction Latency to Red Light | Baseline (Visit 1)
  Maximum pupil constriction to red light will be quantified using chromatic pupillometry with a handheld chromatic pupillometer. Constriction latency is defined as the time from red light onset to the first detectable decrease in pupil diameter relative to baseline. It is measured in seconds.
Post-illumination Pupillary Responses | Baseline (Visit 1)
  Post-illumination pupillary responses (PIPR) will be quantified using chromatic pupillometry with a handheld chromatic pupillometer. PIPR refers to the sustained pupil constriction that persists after the termination of a light stimulus.

SECONDARY OUTCOMES:
Anticipatory Pupil Size | Immediately after the procedure
  Anticipatory pupil size will be assessed using an eyetracker measuring pupil size throughout PVT and oddball tasks. Anticipatory pupil size will be quantified by median pupil size prior stimulus onset.
Hit Rate | Immediately after the procedure
  Hit Rate assessed using a laboratory-based auditory oddball task. Auditory tones will be presented via headphones while participants view a fixation display on a monitor and respond using a keyboard. Hit rate is defined as the proportion of correctly detected target tones relative to the total number of target tones presented during the auditory oddball task.
False Alarm Rate | Immediately after the procedure
  False alarm rate is assessed using a laboratory-based auditory oddball task. Auditory tones will be presented via headphones while participants view a fixation display on a monitor and respond using a keyboard. False alarm rate is quantified as the proportion of responses made to non-target tones relative to the total number of non-target tones presented during the auditory oddball task.
Correct Rejection Rate | Immediately after the procedure
  Correct rejection rate is assessed using a laboratory-based auditory oddball task. Auditory tones will be presented via headphones while participants view a fixation display on a monitor and respond using a keyboard. Correct rejection rate is defined as the proportion of non-target tones for which no response is made (i.e., correctly ignored non-target tones) relative to the total number of non-target tones presented during the auditory oddball task.
Miss Rate | Immediately after the procedure
  Miss rate is assessed using a laboratory-based auditory oddball task. Auditory tones will be presented via headphones while participants view a fixation display on a monitor and respond using a keyboard. Miss rate is quantified as the proportion of target tones for which no response is made (i.e., missed targets) relative to the total number of target tones presented during the auditory oddball task.
Visual Behavior During Time Estimation Task | Immediately after the procedure
  Eye-movement behavior during the time estimation task will be assessed using video-based eye tracking. Metrics will characterize visual behavior during interval estimation and include fixation count and duration, saccade frequency, and related summary measures averaged across trials.
Secondary Risk Taking Metrcis | Immediately after the procedure
  Additional performance metrics from the Balloon Analogue Risk Task (BART) will be derived to further characterize task behavior and outcomes. These metrics include the number of balloon explosions, total earnings accumulated, and related summary measures averaged across trials. These outcomes provide complementary information on risk-reward decision-making beyond the adjusted average pump count.
Reward Seeking Behavior | Immediately after the procedure
  Reward seeking behavior is assessed using the Balloon Analogue Risk Task (BART), a computerized decision-making task. The number of trilas played will be quantified as a metric reflecting reward seeking behavior.
Risk/Reward-Related Visual Behavior | Immediately after the procedure
  Eye-movement behavior during the Balloon Analogue Risk Task (BART) will be assessed using video-based eye tracking. Metrics will characterize visual behavior during decision-making and include areas visited (count and duration), fixation count and duration, saccade frequency, and related summary measures averaged across trials.
Daytime average light levels (lux) | 8-16 days between the visits
  Daytime average light levels (lux) collected using wearable light sensors.
Daytime average melanopic lux | 8-16 days between the visits
  Daytime average melanopic lux collected using wearable light sensors.
Time spent outdoors | 8-16 days between the visits
  Calculated time spent outdoors collected using the wearable light sensors.
Nighttime average melanopic lux | 8-16 days between the visits
  Nighttime average melanopic lux collected using wearable light sensors.
Time spent over 250 or other melanopic EDI threshold during daytime | 8-16 days between visits
  Time spent over 250 or other melanopic EDI threshold during daytime measured using the wearable light sensor
Time spent under 10 or other melanopic EDI threshold during nighttime | 8-16 days between visits
  Time spent below 10 melanopic lux or other thresholds during nighttime measured using the wearable light sensor

CONTACTS AND LOCATIONS:
Overall Officials: Raymond P. Najjar, PhD, Principal Investigator — National University of Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore National Eye Center, Singapore

IPD SHARING:
Plan to Share IPD: No